CLINICAL TRIAL: NCT04989088
Title: Neurofeedback Training to Restore Hemispheric Imbalance in Dyslexia
Brief Title: Neurofeedback Training for Dyslexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Alice Cancer, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NF-DYSL
Record Dates: First submitted 2021-07-15; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Dyslexia; Reading Problem
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left theta/beta and right beta/theta NF training (Experimental)
  Interventions: Device: ProComp5 Infiniti System w/BioGraph Infiniti Software
- Sham NF training (Placebo Comparator)
  Interventions: Device: ProComp5 Infiniti System w/recorded videos

INTERVENTIONS:
Device: ProComp5 Infiniti System w/BioGraph Infiniti Software — Left theta/beta NF training in combination with right beta/theta NF training in temporo-parietal regions, for 40 minutes (with a 20-minute break period)
  Arms: Left theta/beta and right beta/theta NF training
Device: ProComp5 Infiniti System w/recorded videos — Sham NF training using pre-recorded videos, for 40 minutes (with a 20-minute break period)
  Arms: Sham NF training

SUMMARY:
The study aims at testing a Neurofeedback (NF) training specifically designed for inducing a functional hemispheric imbalance of the tempo-parietal regions in individuals with dyslexia. A randomized clinical trial aimed at comparing two experimental conditions is described: a) Left theta/beta NF training in combination with right beta/theta NF training and b) sham NF training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dyslexia or reading performance 2 SD below the norm
* Average intelligence

Exclusion Criteria:

* Psychiatric conditions
* Comorbidity with neurodevelopmental disorders
* Neurological disorders
* Epilepsy
* Enrollment in linguistic or literature university courses

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
EEG recording - ProComp5 Infiniti System | 1 hour
  EEG power in theta/beta band recording in TP7 and TP8
Phonological task (Spironelli & Angrilli, 2006) accuracy | 1 hour
  Computerized rhyme decision task - n. of errors
Phonological task (Spironelli & Angrilli, 2006) speed | 1 hour
  Computerized rhyme decision task - response time (ms)
Semantic task (Spironelli & Angrilli, 2006) speed | 1 hour
  Computerized semantic decision task - response time (ms)
Semantic task (Spironelli & Angrilli, 2006) accuracy | 1 hour
  Computerized semantic decision task - n. of errors
Text reading speed - LSC-SUA Battery (Cornoldi, Montesano & Valenti, 2020) | 1 hour
  Text reading speed measured in syllables / seconds
Text reading accuracy - LSC-SUA Battery (Cornoldi, Montesano & Valenti, 2020) | 1 hour
  Text reading accuracy measured in n. of errors
Word reading speed - LSC-SUA Battery (Cornoldi, Montesano & Valenti, 2020) | 1 hour
  Word reading speed measured in syllables / seconds
Word reading accuracy - LSC-SUA Battery (Cornoldi, Montesano & Valenti, 2020) | 1 hour
  Word reading accuracy measured in n. of errors
Psuedo-word reading speed - LSC-SUA Battery (Cornoldi, Montesano & Valenti, 2020) | 1 hour
  Psuedo-word reading speed in syllables / seconds
Psuedo-word reading accuracy - LSC-SUA Battery (Cornoldi, Montesano & Valenti, 2020) | 1 hour
  Psuedo-word reading accuracy measured in n. of errors

SECONDARY OUTCOMES:
Rapid automatized naming speed (RAN, De Luca, Di Filippo, Judica, Spinelli & Zoccolotti, 2005) | 1 hour
  Rapid automatized naming (RAN) speed measured in seconds
Rapid automatized naming accuracy (RAN, De Luca, Di Filippo, Judica, Spinelli & Zoccolotti, 2005) | 1 hour
  Rapid automatized naming (RAN) accuracy measures in n. of errors
Digit Span (Wechsler Adult Intelligence Scale - Fourth Edition, WAIS-IV) | 1 hour
  Digit forward and digit backword task

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cancer A, Vanutelli ME, Lucchiari C, Antonietti A. Using Neurofeedback to Restore Inter-Hemispheric Imbalance: A Study Protocol for Adults With Dyslexia. Front Psychol. 2021 Nov 5;12:768061. doi: 10.3389/fpsyg.2021.768061. eCollection 2021. PMID 34803851